CLINICAL TRIAL: NCT06074198
Title: Sickle Cell Children's Exercise Study Determining the Effects of a Targeted Exercise Training Program on Neuromuscular Performance, Locomotor Efficiency, and Exercise Tolerance in Children with Sickle Cell Disease.
Brief Title: Sickle Cell Children's Exercise Study (SuCCESs)
Acronym: SuCCESs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, victoria marchese, professor, Chair, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00107858
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Disease
Keywords: physical therapy; neuromotor performance; functional capacity
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: feasibility study
Masking Description: One physical therapist will perform the pre- and post-test assessment measures and another pediatric physical therapist will perform the intervention sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical Therapy Exercise (Experimental): There will be no control group and only one intervention delivered
  Interventions: Behavioral: SuCCESs

INTERVENTIONS:
Behavioral: SuCCESs — strengthening and endurance exercises

SUMMARY:
The Sickle Cell Children's Exercise Study (SuCCESs) will explore the feasibility and effects of a moderate intensity strengthening, balance, speed, and agility intervention program in children with sickle cell disease.

DETAILED DESCRIPTION:
Participants will perform the baseline assessment and after six weeks of performing the SuCCESs program the participants will perform a post-intervention assessment. Participants will be asked to attend a total of six physical therapy in-person sessions (1x/week) at the University of Maryland Department of Physical Therapy and Rehabilitation Science and to perform 12 home program sessions.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-17 years of age diagnosed with sickle cell disease

Exclusion Criteria:

* Diagnosis of neurological disorder, not related to sickle cell disease
* Lower extremity injury such as a fracture with a cast

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
knee extension strength | week 1 and week 7
  dynamometry to measure knee extension strength
Rate of Muscle Activation | week 1 and week 7
  Electromyography used to measure rate of muscle activation
exercise tolerance | week 1 and week 7
  6-Minute Walk Test used to measure exercise tolerance
locomotor efficiency | week 1 and week 7
  oxygen uptake used to measure locomotor efficiency
number of sessions attended | throughout the entire study week 1, weeks 2-6, six weeks of intervention, and week 7
  attendance

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland School of Medicine Dept. of Physical Therapy & Rehabilitation Science, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchese V, Rock K, Harpold A, Salazar A, Williams M, Shipper AG. Physical Impairment and Function in Children and Adolescents With Sickle Cell Disease: A Systematic Review. Arch Phys Med Rehabil. 2022 Jun;103(6):1144-1167.e2. doi: 10.1016/j.apmr.2021.08.022. Epub 2021 Sep 27. PMID 34592159
- [Background] Lanza MB, Rock K, Marchese V, Addison O, Gray VL. Hip Abductor and Adductor Rate of Torque Development and Muscle Activation, but Not Muscle Size, Are Associated With Functional Performance. Front Physiol. 2021 Oct 14;12:744153. doi: 10.3389/fphys.2021.744153. eCollection 2021. PMID 34721067
- [Background] Ho S, Rock K, Marchese V. Diaphragm excursion correlates with performance and ventilation on the 6-min walk test in children with sickle cell disease. Pediatr Pulmonol. 2023 Jun;58(6):1665-1673. doi: 10.1002/ppul.26373. Epub 2023 Mar 8. PMID 36843306
- [Background] Rock K, Nelson C, Addison O, Marchese V. Assessing the Reliability of Handheld Dynamometry and Ultrasonography to Measure Quadriceps Strength and Muscle Thickness in Children, Adolescents, and Young Adults. Phys Occup Ther Pediatr. 2021;41(5):540-554. doi: 10.1080/01942638.2021.1881200. Epub 2021 Feb 9. PMID 33563044